CLINICAL TRIAL: NCT05399810
Title: Effects of Computer Application (ICOGNI) Based Training Along With Routine Physical Therapy on Executive Functions and Motor Skills in Cerebral Palsy
Brief Title: Computer Application (ICOGNI) Based Training Along With Routine Physical Therapy on Executive Functions and Motor Skills in Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/1001/2021
Record Dates: First submitted 2022-02-12; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-02

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer Application (ICOGNI) Training (Experimental): Apart from routine physical therapy, participants in this group will be randomized to active training after baseline assessment. Participants will be given App-based training which will include multiple games with multiple levels along with routine physiotherapy. The active group will start training immediately and will have 8 weeks to perform the 40 training sessions.
  Interventions: Other: Computer Application (ICOGNI) Training
- Conventional group (No Intervention): Participants in are already being given routine physiotherapy which includes range of motion exercises, stretching and strengthening exercises of upper extremity, fine motor activities, functional activities, and cognitive activities (art and crafts, placing objects in specific positions, organizing objects, color sorting games, teamwork, and moving and tracing objects).

INTERVENTIONS:
Other: Computer Application (ICOGNI) Training — Participants will be given App-based training under supervision for 40 sessions, which will include multiple games with multiple levels along with routine physiotherapy.
  Arms: Computer Application (ICOGNI) Training

SUMMARY:
This study design will be randomized controlled trial. Subjects will be selected for data collection from the Physiotherapy Department, Institute of Pediatric and Rehabilitation of The University of Lahore Teaching Hospital and Central Park Teaching Hospital, Lahore. Subjects will be randomly allocated into two equal groups, conventional group (group A) and an experimental group (group B). Conventional group will be receiving routine physical therapy and Experimental group will be receiving Computer application-based training and routine physical therapy. Pre and post intervention data will be taken from Gross Motor Function Classification System, Manual Ability Classification System, Mini-Mental State Examination for Children and Quality of Upper Extremity Skills Test for data analysis.

DETAILED DESCRIPTION:
This study design will be randomized controlled trial. Subjects will be selected for data collection from the Physiotherapy Department, Institute of Pediatric and Rehabilitation of The University of Lahore Teaching Hospital and Central Park Teaching Hospital, Lahore. Subjects will be randomly allocated into two equal groups, conventional group (group A) and an experimental group (group B). Conventional group will be receiving routine physical therapy and an Experimental group will be receiving Computer application-based training and routine physical therapy. Training will be given once a day, five times a week for total 8 weeks. For conventional group, the training duration for each session will be 30 minutes with 5 minutes of rest period and for experimental group, 60 minutes with 10 minutes of rest period in between. Participants in conventional group will be given routine physiotherapy which will include range of motion exercises, stretching and strengthening exercises of upper extremity, fine motor activities, functional activities, and cognitive activities (art and crafts, placing objects in specific positions, organizing objects, color sorting games, teamwork, and moving and tracing objects). Participants in experimental group will be given routine physiotherapy along with App-based training. The routine physiotherapy will be the same as given to the control group and app-based training will include multiple games with multiple levels. Pre and post intervention data will be taken from Gross Motor Function Classification System, Manual Ability Classification System, Mini-Mental State Examination for Children and Quality of Upper Extremity Skills Test for data analysis. For the assessment of executive function skills, Mini-mental State Examination For Children (MMC) will be used and for motor skills, Quality Of Upper Extremity Skills Test (QUEST) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 8-16 years.
* Children with diagnosed spastic unilateral CP
* Who are able to follow instructions
* Respond to visual and auditory stimuli
* Who are able to handle computer/ tablet
* School going children
* One of the parents should be literate
* MMC score less than 24 (mild to moderate impairment)
* GMFCS level 2

Exclusion Criteria:

* Presence of epilepsy
* Complex communication disorders
* Any surgical procedure

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination for Children (MMC) | 8 weeks
  Mini-Mental State Examination for Children (MMC) is an adapted version of the Mini-Mental State Examination. The Mini-Mental Examination for Children(MMC) is a widely used tool for assessing global cognitive deficits with a maximum score of 37.
Quality of Upper Extremity Skills Test (QUEST) | 8 weeks
  Quality of Upper Extremity Skills Test (QUEST) is a reliable measure of gross motor upper limb functions in children with CP. This measure assesses mainly four domains: dissociated movement, grasp, protective extension, and weight bearing.

CONTACTS AND LOCATIONS:
Overall Officials: Hadeeqa Momin, MSPTN*, Principal Investigator — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pirila S, van der Meere JJ, Rantanen K, Jokiluoma M, Eriksson K. Executive functions in youth with spastic cerebral palsy. J Child Neurol. 2011 Jul;26(7):817-21. doi: 10.1177/0883073810392584. Epub 2011 Mar 11. PMID 21398561
- [Background] Boyd RN, Baque E, Piovesana A, Ross S, Ziviani J, Sakzewski L, Barber L, Lloyd O, McKinlay L, Whittingham K, Smith AC, Rose S, Fiori S, Cunnington R, Ware R, Lewis M, Comans TA, Scuffham PA. Mitii ABI: study protocol of a randomised controlled trial of a web-based multi-modal training program for children and adolescents with an Acquired Brain Injury (ABI). BMC Neurol. 2015 Aug 19;15:140. doi: 10.1186/s12883-015-0381-6. PMID 26286324